CLINICAL TRIAL: NCT00485719
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL765 Administered Orally Daily to Subjects With Solid Tumors
Brief Title: Study of the Safety and Pharmacokinetics of XL765 (SAR245409) in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11440; 2007-002437-36 (EudraCT Number); XL765-001 (Other: (other study code))
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Cancer
Keywords: Cancer; Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — XL765

ARMS (2):
- 1 (Experimental): Twice daily (bid) dosing
  Interventions: Drug: XL765 (SAR245409)
- 2 (Experimental): Once daily (qd) dosing
  Interventions: Drug: XL765 (SAR245409)

INTERVENTIONS:
Drug: XL765 (SAR245409) — Gelatin capsules supplied in 5-mg, 10-mg, and 50-mg strengths administered orally

SUMMARY:
The purpose of this study is to determine the safety and tolerability of XL765. XL765 is a new chemical entity that inhibits the kinases PI3K and mTOR. In preclinical studies, inactivation of PI3K has been shown to inhibit growth and induce apoptosis (programmed cell death) in tumor cells, whereas inactivation of mTOR has been shown to inhibit the growth of tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologically confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective, and there are no therapies known to prolong survival.
* The subject has disease that is assessable by tumor marker, physical, or radiologic means.
* The subject is at least 18 years old.
* The subject's weight is at lease 40 kg.
* The subject has an Eastern Cooperative Oncology Group performance status of 0 - 2.
* The subject has adequate organ and bone marrow function.
* The subject has fasting plasma glucose < 120 mg/dL at screening.
* for subjects who are to be enrolled into the Expanded MTD Cohort and Lower-Dose Tumor Genetic Alteration Subjects:

  1. tumor tissue amenable to serial biopsy;
  2. additional informed consent
* The subject is capable of understanding the protocol and has signed the informed consent.
* Sexually active subjects (male and female) must use medically acceptable methods of contraception during the course of the study.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening.
* If the subject has received more than 3 prior regimens of cytotoxic chemotherapy, more than 2 biologic regimens, or more than 3000 cGy to >25% of his or her bone marrow, the sponsor must determine subject suitability before enrollment.
* The subject has had no other diagnosis of malignancy (unless non-melanoma skin cancer, in situ carcinoma of the cervix, or a malignancy diagnosed ≥ 2 years ago, and has had no evidence of disease for 2 years prior to screening for this study.)

Exclusion Criteria:

* The subject has received anticancer treatment (chemotherapy, radiotherapy, cytokines, or hormones) within 30 days (6 weeks for nitrosoureas, mitomycin C, or bicalutamide) before the first dose of XL765.
* The subject has received radiation to > 25% of his or her bone marrow.
* The subject has not recovered from adverse events, except Grade 2 alopecia, due to other investigational or other agents administered prior to study enrollment.
* The subject has received another investigational agent within 30 days or the first dose of XL765 or a small-molecule kinase inhibitor within 14 days or 5 half-lives.
* The subject is known to have diabetes
* The subject has uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* The subject has psychiatric illness/social situation that would limit compliance with study requirements.
* The subject is pregnant or breast feeding.
* The subject is known to be positive for HIV.
* The subject has a known allergy or hypersensitivity to components of the XL765 formulation.
* The subject has a baseline corrected QT interval > 450 ms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose (MTD) of daily oral administration of XL765 in two treatment schedules | Assessed at each visit/periodic visits

SECONDARY OUTCOMES:
Plasma pharmacokinetics of daily oral administration of XL765 in two treatment schedules | Assessed at periodic visits
Pharmacodynamic effects of XL765 on tumor tissue when administered at the MTD in two treatment schedules | Assessed during periodic vixits after MTD is determined

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (3):
  - Investigational Site Number 1302, Detroit, Michigan
  - Investigational Site Number 1435, Omaha, Nebraska
  - Investigational Site Number 1402, San Antonio, Texas
- Investigational Site Number 3411, Barcelona, Spain